CLINICAL TRIAL: NCT06484192
Title: Randomized Controlled Trial of Postoperative Inpatient Ketorolac and Outpatient Naproxen Use Following Elective Lumbar Spine Fusion
Brief Title: Pain Control After Lumbar Spine Fusion
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CKEP2024.0800
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Spine Fusion; NSAID (Non-Steroidal Anti-Inflammatory Drug); Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Naproxen; Ketorolac; Oxycodone; Tablets; metaxalone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1: NSAID Group (Active Comparator): Participants in the NSAID group will receive NSAIDs in addition to our standard postoperative regimen after their Lumbar spine fusion surgery
  Interventions: Drug: Naproxen 500 Mg; Drug: Ketorolac; Drug: OxyCODONE 5 mg Oral Tablet; Drug: Metaxalone 800 MG
- Group 2: Control Group (Active Comparator): Participants in the control group will only receive our standard postoperative regimen after their Lumbar spine fusion surgery
  Interventions: Drug: OxyCODONE 5 mg Oral Tablet; Drug: Metaxalone 800 MG

INTERVENTIONS:
Drug: Naproxen 500 Mg — participants will receive Naproxen (500 mg) to take for 7 days after surgery as needed
  Arms: Group 1: NSAID Group
Drug: Ketorolac — participants will receive Ketorolac (15 mg) immediately after surgery
  Arms: Group 1: NSAID Group
Drug: OxyCODONE 5 mg Oral Tablet — participants will receive OxyCODONE (5 mg) to take for 7 days after surgery as needed
Drug: Metaxalone 800 MG — participants will receive Metaxalone (800 MG) to take for 7 days after surgery as needed

SUMMARY:
The purpose of this randomized controlled trial is to determine if patients who receive non-steroidal anti-inflammatory medications (NSAIDs) following elective lumbar spinal fusion have increased rates of symptomatic nonunion requiring revision spinal surgery at two-years follow-up, compared to those who do not receive NSAIDs.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age, ≥1-level planned lumbar spinal fusion
* Capacity to enroll
* English speaking

Exclusion Criteria:

* Chronic kidney disease (preoperative creatinine ≥1.4)
* History of gastrointestinal bleed or peptic ulcer disease
* History of spinal fusion nonunion
* Non-steroidal anti-inflammatory drug allergy
* Previously diagnosed coagulopathy
* Preoperative thrombocytopenia (platelets <100,000)
* Connective tissue disease
* Operative indication due to infection, neoplasm, or trauma
* Currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 428 (Estimated)
Dates: Start 2024-06-28 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Fusion failure | 2 years
  Failure of fusion surgery will be measured by the rate of revisions as demonstrated by participant x-rays

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States